CLINICAL TRIAL: NCT03026452
Title: Effectivity and Safety of Ultrasound-guided Percutaneously Radiofrequency Ablation for Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFA-001
Record Dates: First submitted 2017-01-04; First posted 2017-01-20 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2016-12

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

ARMS (1):
- RFA(radiofrequency ablation) (Experimental): The investigators used percutaneously US-guided RFA(radiofrequency ablation) for small hepatocellular carcinoma,and estimated the safety and efficacy of this treatment through 2-year follow-up of US/CEUS/CT/MRI and the tumor markers.
  Interventions: Procedure: US-guided RFA

INTERVENTIONS:
Procedure: US-guided RFA — The investigators used percutaneously US-guided radiofrequency ablation for patients with small hepatocellular carcinoma,and estimated the safety and efficacy of this treatment through 2-year follow-up of US/CEUS/CT/MRI and the tumor markers.

SUMMARY:
To evaluate the safety and efficacy of ultrasonography (US) -guided radiofrequency ablation for liver tumors, the investigators used preoperative and postoperative US/CEUS(contrast-enhanced ultrasonography)/CT/MRI to assess lesions, and laboratory tests including the tumor markers to evaluate the general condition of patients. Intraoperative US/CEUS/CT would be applied to monitor ablation lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with small hepatocellular carcinoma (single or multiple nodules of less than 3 cm in diameter), Patients with Child-Pugh A/B, Patients with PLT(platelet count) ≥ 50*10e9/L and PT(prothrombin time) ≤ 20s.

Exclusion Criteria:

* Patients with blood coagulation dysfunction, ChildPugh score≥3, severe cardiopulmonary disease, intolerant anesthesia and upper gastrointestinal bleeding in shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Tumor size assessed by MRI | through study completion, an average of 2 year
  Tumor size was estimated by MRI.

SECONDARY OUTCOMES:
Carcinoembryonic Antigen (CEA) level assessed by ELISA | through study completion, an average of 2 year
  CEA level was assessed by enzyme linked immunosorbent assay (ELISA).
Alpha Fetoprotein (AFP) level assessed by ELISA | through study completion, an average of 2 year
  AFP level was assessed by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Sasaki K, Margonis GA, Andreatos N, Kim Y, Wilson A, Gani F, Amini N, Pawlik TM. Combined resection and RFA in colorectal liver metastases: stratification of long-term outcomes. J Surg Res. 2016 Nov;206(1):182-189. doi: 10.1016/j.jss.2016.06.098. Epub 2016 Jul 4. PMID 27916360
- [Result] Giorgio A, Merola MG, Montesarchio L, Merola F, Santoro B, Coppola C, Gatti P, Amendola F, DI Sarno A, Calvanese A, Matteucci P, Giorgio V. Sorafenib Combined with Radio-frequency Ablation Compared with Sorafenib Alone in Treatment of Hepatocellular Carcinoma Invading Portal Vein: A Western Randomized Controlled Trial. Anticancer Res. 2016 Nov;36(11):6179-6183. doi: 10.21873/anticanres.11211. PMID 27793949
- [Result] Makino Y, Imai Y, Igura T, Kogita S, Sawai Y, Fukuda K, Iwamoto T, Okabe J, Takamura M, Fujita N, Hori M, Takehara T, Kudo M, Murakami T. Feasibility of Extracted-Overlay Fusion Imaging for Intraoperative Treatment Evaluation of Radiofrequency Ablation for Hepatocellular Carcinoma. Liver Cancer. 2016 Oct;5(4):269-279. doi: 10.1159/000449338. Epub 2016 Sep 14. PMID 27781199
- [Result] Aissou S, Cartier V, Hamy A, Plumereau F, Aube C, Lermite E. Radiofrequency in the Management of Colorectal Liver Metastases: A 10-Year Experience at a Single Center. Surg Technol Int. 2016 Oct 26;29:99-105. PMID 27780345
- [Result] Barat M, Fohlen A, Cassinotto C, Jannot AS, Dautry R, Pelage JP, Boudiaf M, Pocard M, Eveno C, Taouli B, Soyer P, Dohan A. One-month apparent diffusion coefficient correlates with response to radiofrequency ablation of hepatocellular carcinoma. J Magn Reson Imaging. 2017 Jun;45(6):1648-1658. doi: 10.1002/jmri.25521. Epub 2016 Oct 20. PMID 27766709
- [Result] Seror O, N'Kontchou G, Nault JC, Rabahi Y, Nahon P, Ganne-Carrie N, Grando V, Zentar N, Beaugrand M, Trinchet JC, Diallo A, Sellier N. Hepatocellular Carcinoma within Milan Criteria: No-Touch Multibipolar Radiofrequency Ablation for Treatment-Long-term Results. Radiology. 2016 Aug;280(2):611-21. doi: 10.1148/radiol.2016150743. Epub 2016 Mar 24. PMID 27010381